CLINICAL TRIAL: NCT06767163
Title: Development and Applications of Daily-use Fall Risk Assessment Device to Prevent Elderly People from Falling
Brief Title: Developing a Daily-use Fall Risk Assessment Device in Clinical Setting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority Hong Kong West Cluster (Unknown)
Responsible Party: Principal Investigator, Prof. Xi Ning, Head of Department; Chair Professor of Robotics and Automation; Director of Advanced Technologies Institute, The University of Hong Kong, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: UW 24-540
Record Dates: First submitted 2025-01-06; First posted 2025-01-09 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Falls; Balance Assessment
Keywords: Fall prevention; Older adults; Balance ability assessement systems; Sensor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group (Experimental): Older adults with zero time of falls in the past twelve months will be treated as the reference group. Older adults with at least one time of falls in the past twelve months will use the device to assess their balance ability by attending three rounds of the tests.
  Interventions: Device: iBalance

INTERVENTIONS:
Device: iBalance — Participants will engage in the device test, clinical assessment tests. The whole test will last twelve months, and the outcome will be assessed pre- and post-implementation for comparison and validation.
  The intervention results are used to compared with traditional tests and clinical diagnosis, to identify whether the sensor provides a higher accuracy in predicting fall risk, and to explore the feasibility of the sensor in clinical scenarios.

SUMMARY:
Study Objectives Objective 1: Compare the fall risk assessment results between balance sensors, traditional tests, and clinical diagnoses.

Objective 2: Improve the feasibility of using sensors to assess fall risk among older patients in the hospital.

The investigators select Hong Kong as the region for the experiment. Specifically, the community clinics and daytime hospitals are the actual onsite locations for experimenting. The specific venues of these locations need an electrical power supply and a flat ground for conducting the device test. Patients will be recruited for the development and testing of a device for fall risk assessment, study participants will be involved in balancing assessments, and questionnaire surveys, their medical records will be accessed. And during these tests and questionnaire surveys, the investigators will take photos, videos, and or audio recordings.

ELIGIBILITY:
Inclusion Criteria:

1. Older adults aged 60 years and above;
2. Understand Cantonese or Mandarin or English;
3. Clinical patients in the clinics.

Exclusion Criteria:

1. Unable to give written informed consent (e.g., illiterate or with cognitive impairment);
2. Inability to stand for 30 seconds without any assistance.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Precision assessment of falling risk prediction | six months
  A primary outcome is the precision assessment of falling risk prediction both from device and clinical diagnose.
  The specific measurement variables for this primary outcome are the classification results of high/low falling risk based on the results (a composite result) of the device test and participants' actual falling incident indicators, including the number of falls, the severity of falling incidents after the device test, and medical history of the participants (eg. the history of the emergency, surgery, and diagnosed disease in the past three years), as well as the diagnosis results of the fall risk by clinical professionals. These results can be shown through the sensitivity and specificity analysis of the device evaluation.

SECONDARY OUTCOMES:
Feasibility of fall risk assessment by using balance sensor in clinical settings | six months
  The secondary outcome is the specific fall risk results given by the device and the participant's body data measurement, demographic information, and survey data about user experience and adoption.
  Additionally, the ideas from clinical professionals on the better application of the device in hospitals will also be regarded as the secondary outcome of this study.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data collected in this study will be published and submitted to academic journals to share with other researchers.
Supporting Information: Study Protocol
Time Frame: No limitations on the publications
Access Criteria: No limitations on the publications